CLINICAL TRIAL: NCT03345160
Title: Open Label Peanut Oral Immunotherapy in Children: IMPACT Follow Up Study
Brief Title: Peanut Oral Immunotherapy in Children: IMPACT Follow Up Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00150453
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Treatment Efficacy

STUDY DESIGN:
Intervention Model Description: Open Label crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peanut Flour: Open label peanut OIT (Experimental): This is an open label treatment for subjects who had previously received placebo treatment in a prior peanut OIT study
  Interventions: Drug: Peanut Flour

INTERVENTIONS:
Drug: Peanut Flour — open label oral immunotherapy
  Other Names: Peanut Oral Immunotherapy

SUMMARY:
This application is being submitted as a follow-up to Protocol "Oral Immunotherapy for Induction of Tolerance in Peanut Allergic Children-The IMPACT Study." The IMPACT study was a double-blind, placebo-controlled study of peanut oral immunotherapy in children 12-48 months of age. As part this protocol, all participants who received placebo treatment were promised the opportunity to receive open label treatment at the conclusion of the double-blind phase and initial follow-up. At the time of submitting that protocol, the investigator did not specify any detailed protocol for the open label crossover treatment, as this is an evolving field, but the investigator is now ready to offer this open label treatment as promised.

DETAILED DESCRIPTION:
This study will enroll up to 20 subjects aged 4-9 years old who were enrolled in the placebo arm of the IMPACT study.

Once subjects have completed participation in the IMPACT study, subjects will be offered the option of participating in this open label, peanut oral immunotherapy study.

After the informed consent has been signed, subjects will undergo an initial dose escalation to peanut protein to establish the starting dose for the build-up phase. The starting dose of peanut protein for the build-up phase will be the highest tolerated dose during the initial dose escalation. The subject will return to the study site and the first starting dose of peanut protein will be given under observation. Subjects will be sent home with doses of peanut protein to administer at home.

Subject will return every 2 weeks for dose adjustments. Once subjects have tolerated a dose under observation, subjects will then continue dosing at home with OIT and return to the research unit every 2 weeks for a 1-step dose escalation to a maximum daily dose of 1000 mg. Participants who do not reach the 1000mg dose by 40-weeks of build-up phase may enter the maintenance phase at their highest tolerated dose.

When subjects reach their maximum tolerated dose of either 1000 mg per day, or the maximum tolerated dose during the 40 weeks of the build-up phase, subjects will enter the maintenance phase. Subjects will continue daily dosing of peanut protein at the maximum tolerated dose during the 12-week maintenance phase.

At the end of the maintenance phase, subjects will undergo an open peanut oral food challenge to a maximum of 4000 mg of peanut protein to determine individualized guidelines for the introduction of peanut into the subject's diet based on the outcome of the open peanut challenge The primary objective of this protocol is to provide open label peanut oral immunotherapy (OIT) for those subjects who received placebo treatment in the IMPACT Study .

Secondary objectives will include:

1. Efficacy of the treatment, as defined by an end of treatment oral peanut challenge.

Safety, as measured by the incidence of adverse events and the proportion of subjects who discontinue treatment due to adverse events

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for enrollment as study participants, including participants who:

* Subjects who were randomized to the placebo arm of protocol NA_00077852 "Oral Immunotherapy for Induction of Tolerance in Peanut Allergic Children."
* Parent guardian must be able to understand and provide informed consent
* Peanut allergy, as defined by a reaction to a cumulative dose of ≤1000 mg of peanut protein during the End-of-Treatment food challenge from Protocol NA_00077852 "Oral Immunotherapy for Induction of Tolerance in Peanut Allergic Children"

Exclusion Criteria:

Patients who meet any of these criteria are not eligible for enrollment as study participants, including participants who:

* Inability or unwillingness of a parent guardian to give written informed consent or comply with study protocol
* History of severe anaphylaxis to peanut, defined by severe hypoxia, hypotension, neurological compromise, confusion, cardiovascular collapse, or loss of consciousness
* Significant chronic disease (other than asthma, rhinitis, or atopic dermatitis) requiring therapy; e.g., heart disease or cystic fibrosis which is judged by the investigator to have potential impact on study outcomes or safety.
* Severe or poorly controlled atopic dermatitis per investigator's discretion
* Past or current history of eosinophilic gastrointestinal disease
* Diagnosis of asthma that meets any of the following criteria:

  * Uncontrolled asthma (as per Global Initiative for Asthma [GINA] latest guidelines)
  * History of 2 or more systemic corticosteroid courses or 1 systemic course within the 3 previous months prior to visit 1 for treating wheezing
  * Prior intubation/mechanical ventilation for asthma
* Currently receiving β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy.
* Current participation in another clinical trial or participation in another clinical trial in the last 90 days

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Derived] Kanchan K, Cerosaletti K, Perry JA, DuToit G, Manohar M, Ling H, Paschall JE, Sanda S, Chinthrajah RS, Nepom GT, Nadeau KC, Jones SM, Lack G, Ruczinski I, Mathias RA. Genetic Determinants of Peanut-Specific IgG4 Levels in the Context of Sustained Oral Peanut Exposure in the LEAP Study. Immunology. 2026 Jan 30. doi: 10.1111/imm.70098. Online ahead of print. PMID 41615410
- [Derived] Jones SM, Kim EH, Nadeau KC, Nowak-Wegrzyn A, Wood RA, Sampson HA, Scurlock AM, Chinthrajah S, Wang J, Pesek RD, Sindher SB, Kulis M, Johnson J, Spain K, Babineau DC, Chin H, Laurienzo-Panza J, Yan R, Larson D, Qin T, Whitehouse D, Sever ML, Sanda S, Plaut M, Wheatley LM, Burks AW; Immune Tolerance Network. Efficacy and safety of oral immunotherapy in children aged 1-3 years with peanut allergy (the Immune Tolerance Network IMPACT trial): a randomised placebo-controlled study. Lancet. 2022 Jan 22;399(10322):359-371. doi: 10.1016/S0140-6736(21)02390-4. PMID 35065784

RESULTS

PARTICIPANT FLOW:
Groups:
- Peanut Flour: Open Label Peanut OIT: This is an open label treatment for subjects who had previously received placebo treatment in a prior peanut oral immunotherapy (OIT) study
  Peanut Flour: open label oral immunotherapy
Period: Overall Study
Arm/Group | Peanut Flour: Open Label Peanut OIT
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Peanut Flour: Open Label Peanut OIT
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.6 [6 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: Number of participants who reported symptoms which were collected as AEs using CTCAE v4.0.
Time Frame: up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Flour: Open Label Peanut OIT
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Amount of Peanut Protein Tolerated at the End-of-treatment Peanut Challenge
Description: This measure assessed the amount of peanut protein [in milligrams (mg)] tolerated by each participant at the end-of-treatment peanut challenge.
Time Frame: up to 52 weeks
Population: Data reported for each participant.
Measure: Number; unit: mg
Arm/Group | Peanut Flour: Open Label Peanut OIT
Number analyzed (Participants) | 7
mg
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 4000
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 4000
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 4000
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 4000
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 4000
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 4000
  Participant 7: number analyzed (Participants) | 1
  Participant 7 | 2000

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: All 7 subjects reported mild symptoms with at least one IP administration. These reactions were collected and reported as AEs. These allergic reactions were expected.
Arm/Group | Peanut Flour: Open Label Peanut OIT
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peanut Flour: Open Label Peanut OIT (N=7)
Mild allergic reaction-Initial Dose Escalation (General disorders) | 4 (4)
Mild allergic reaction-Dosing related (General disorders) | 7 (158)
Gastroenteritis (Gastrointestinal disorders) | 1 (3)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (5)
influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Otitis Media (Ear and labyrinth disorders) | 3 (3)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Allergic Conjunctivitis (Eye disorders) | 1 (1)
Eczema Flare (Skin and subcutaneous tissue disorders) | 2 (4)
Vomiting-not associated with dosing (Gastrointestinal disorders) | 3 (4)
Strept Throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea-not associated with dosing (General disorders) | 2 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic Reaction -not related to dosing (General disorders) | 1 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Otitis Externa (Ear and labyrinth disorders) | 1 (1)
Back pain-related to a fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash-not related to dosing (Skin and subcutaneous tissue disorders) | 1 (2)
Dehydration (General disorders) | 1 (1)
GERD-not related to dosing (Gastrointestinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03345160/Prot_SAP_000.pdf